CLINICAL TRIAL: NCT02930148
Title: Personalised Guidance Service for Lifestyle Management and Obesity Prevention in Teen-agers: A Multicenter Quasi-experimental Pilot Study
Brief Title: Personalised Guidance Service for Lifestyle Management and Obesity Prevention in Teen-agers Pilot Study
Acronym: PEGASO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Agència de Qualitat i Avaluació Sanitàries (Other Government)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); Politecnico di Milano (Other); University of Nottingham (Other); University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 750-PEGASO
Record Dates: First submitted 2016-10-04; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-09

CONDITIONS: Lifestyles
Keywords: mHealth; adolescents; quasi-experimental study; apps; lifestyles; lifestyles knowledge; dietary behaviour; physical activity; sleeping behaviour
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants will be provided with a smart phone (android, version 5.0), two smart garments, a smart garment sensor and an activity bracelet will be provided at month 2 (to minimise the burden on the schools and participants allocating time and resources). The smart phones will have all apps of the PEGASO ecosystem installed.
  Interventions: Other: PEGASO System (ICT based system/mHealth solution)
- Comparative (No Intervention): Participants will be asked to continue their routine daily physical and educational activities related to leading a healthy lifestyle.

INTERVENTIONS:
Other: PEGASO System (ICT based system/mHealth solution) — Participants will be provided with a smart phone with the PEGASO system and will be asked to join the PEGASO community through the PEGASO Portal. Two smart garments, and two sensors will be provided at month 2 (to minimise the burden on the schools and participants allocating time and resources). The PEGASO System allows empowering the participants toward healthy habits, recording what he or she eats, monitor physical activity variables. The serious game is a central motivational component of PEGASO: it has an "energy bar", used up by the player's actions, and replenished when achieving their behavioural goals, and it implements "research" mechanics that require the player to apply and develop their nutritional knowledge. The Bridge allows the connection between the PEGASO ecosystem and the personal health folder by creating a report to be shared with physicians
  Arms: Intervention

SUMMARY:
the aims of the present study is to test the PEGASO system in real life conditions in Lombardy (Italy), England and Scotland (UK) and Catalonia (Spain), as well as to assess changes in teen-agers' awareness and lifestyles after the use of PEGASO system. Specifically, the investigators aim to:

1. To test the usability of PEGASO platform
2. To pilot approaches to testing the effectiveness of the system to:

   1. Evaluate the increase of knowledge/awareness about healthy habits
   2. Assess behavioural change in lifestyle, and specifically on target behaviours In particular, the pilot study will help to assess likely recruitment and retention in a controlled trial, to test the acceptability and utility of assessment procedures, to obtain estimates of effect size and variability to power a future substantive study

DETAILED DESCRIPTION:
A multi-centre quasi experimental controlled pilot study will be undertaken to evaluate a 6 months ICT based intervention, the PEGASO System, to promote healthy habits among adolescents. The study will include adolescents from four sites: England (UK), Scotland (UK), Lombardy (Italy) and Catalonia (Spain). Participants in he intervention group will test the PEGASO ecosystem from October 2016 to March 2017 while those in the comparative group will not have access to the PEGASO ecosystem. The sample selection will be carried out in two stages: in the first phase, schools with medium-low socioeconomic level will be selected by convenience sampling; in the second phase classes will be selected for participation in each school in agreement with schools principals/ head teachers. A total of 525 adolescents from participating high schools will be asked to participate in the study as intervention or comparative group, in a 2:1 ratio. Consequently, approximately, 350 participants of the four pilot sites will be testing the PEGASO platform, whilst 175 will be the comparative group. Decisions about appropriate sample sizes were underpinned by a range of considerations, including the study's aims, operational constraints, the accuracy of the survey estimates and costs.

The PEGASO system is based on the comprehensive Behavior Change Wheel (BCW) framework and in particular by the Capability-Opportunity-Motivation-Behavior (COM-B) system. This provided the theoretical grounding for the content and implementation approach of the behavior change interventions embedded within the components of the PEGASO system. The innovative key component of the PEGASO system is the behavior recognition system which allows detection and evaluation of participants' real-time behavior (collected through other components of the PEGASO system). While the target behaviors allow focusing the intervention on a specific task for each participant, the link between behavior change theory (Behavior Change wheel) and the target behaviors is ensured via the COM-B questionnaire. Participants will have the opportunity to choose one target behavior at the time. When selecting a novel target behavior, participants will be asked to complete the COM-B questionnaire. The answers for each question subset will guide which component of the COM-B behavior system adopt to target the content of the behavior change intervention. For instance, the messaging framework in the PEGASO Companion App will select messages that are associated with participants' preferences expressed in the COM-B questionnaire. This will provide an intervention that is personalized to the different needs of the individual intervention participant.

To analyze the effectiveness of the platform in modifying knowledge/awareness and behaviors the investigators will compare intervention and control groups by utilizing an intention-to-treat (ITT) approach, thus inferring the effect independently from drop-outs and non-adherence.

The participants will be provided with a smart phone (android, version 5.0) for the duration of the study. Two smart garments, a smart garment sensor and an activity bracelet will be provided at month 3. The smart phones will have all apps of the PEGASO ecosystem installed. In addition, participants will be asked to join the PEGASO community by signing in to the PEGASO Portal (http://portal.PEGASOf4f.eu/web/others/sign-in).

PEGASO comprises seven different apps. The objective of the PEGASO Companion app is to encompass the other six apps and provide a seamless and unique experience to the participant. Companion App. The aim of the Companion App is to make active life more attractive, helps participants to eat more healthily and connects participants with their peers. Developed as native Android application (client + server), the Companion is a Personal Digital "Friend" acting as a daily-life guide for coaching, caring for, and empowering the participants in their activities toward healthy habits. The Companion App will allow the user to have dynamic stream of information (about their achievements and the achievements of the other users that chose to connect with the user within the PEGASO system) and to access all other applications. Data acquired via sensors (embedded in the Smartphone or garments) will be presented to the user via a specific interface developed inside the Health Companion App. The Companion App also includes a rewarding system and the gamification module will allow the system to: achieve One time rewards, achieve Cyclic events and achieve Rewards (e.g., fit coins, badges, experience points) for the selected target behavior (diet or physical activity). Challenges app. The Companion app includes a "challenge" component which participants can use for creating and accepting different type of challenges. This application allows users to challenge themselves and other users in a competitive or collaborative way. eDiary app. The eDiary is an application that allows the participant to enter some information about their diet and provides feedback about the healthy eating habit. This app will also provide suggestions (e.g., food groups and recipes) to the user to improve the dietary habits. The eDiary app is gamified in order to improve the participants' experience and to introduce an element of fun that can sustain engagement with the app and eating habits. PEGASO City app. The PEGASO City is a bridge between the digital world of the PEGASO system with the physical world. The app has a twofold role inside the PEGASO Health Companion: firstly, PEGASO City helps teenagers to find places that are part of the PEGASO Stakeholder Ecosystem, and that provide them opportunities to act healthy and progress towards the reach of their target behavior. Secondly, through the empowerment provided by the integration of some of the HealthSquare functionalities, the application provides the teenagers a set of possible interactions and actions that contribute to the gamification process and the rewarding system. Dashboard app. The Dashboard is an application that allows to see all the data acquired by the PEGASO system. The app shows all the activities data such as steps and minutes of activities, sleep time, type of activities made during the course of the day; in addition, it reports if the user reaches the target behavior and awards him/her with badges and trophies. Thanks to the Dashboard the participants are able to check their behavior and perform reflection and self-monitoring by extracting suggestions from the apps. Users can also control the battery and memory status of each PEGASO device. Smart Garments and bracelets sensors. Smart garments consist of a t-shirt/crop top with embedded textile electrodes. The t-shirt/crop top comes with a data logger (monitoring/recording system) which snaps on the front side of the t-shirt by using standard snap buttons. The smart garments measure heart rate (ECG) and physical activities (accelerometer) whereas the bracelet monitors physical activities and sleep. Data collected through garments and bracelets are transferred to a smart phone and linked to the Health Companion app as well as the serious game. Participants will be provided with a User Manual in local languages. Serious game. The game serves a central role as the motivational component of PEGASO. As such, it needs to entertain and engage the player, whilst utilizing the PEGASO ecosystem to capture information about lifestyles and encourage positive health behavior changes. There are two central behavioral mechanisms within the game: a) an "energy bar", used up by the player's actions in the game, and replenished by them achieving their behavioral goals such as increased physical activity or improved diet, and b) the game implements "research" mechanics that require the player to apply and develop their nutritional knowledge of various food sources. The current game format is an infinite game which, through the energy mechanic, promotes regular use and goal-achievement within the PEGASO ecosystem, as well as being conducive to short, frequent play rather than long single sessions. PEGASO Web Portal. The PEGASO Web Portal allows participants to socially interact and learn via training module; two (technological): aggregate data and services across the whole PEGASO platform (images, video, blog materials, activities data, no. of steps, no. of km). Potentially users of the PEGASO Portal are teenagers, parents and experts. The Web portal is accessible from both mobile devices and computers. Report App. The connection between the PEGASO ecosystem and the personal health folder is established through the BRIDGE system and will be deployed and tested in two pilot sites only: namely Lombardy region and Catalonia. The BRIDGE allows extracting health data collected and elaborated into the PEGASO ecosystem and to create a report to be shared with physicians into the personal health folder (PHF).

Chi-squared test will be used to analyze the association between independent qualitative variables, along with the McNemar test for paired samples. The Student t-test will be used for the comparison of means between two groups, and the paired t-test will be applied to assess changes within one same group. Alternatively, the corresponding nonparametric tests will be used, as required. The relationship between quantitative variables will be analyzed using Pearson's correlation coefficient or Spearman coefficient in the case of asymmetrically distributed variables. Multivariate linear regression analysis and logistic regression analysis will be used to analyze the variables determining the changes in physical activity and eating and sleeping habits. In order to analyze the effect of the intervention, comparison will be made of the changes observed in the comparison group (CG) versus the intervention group (IG), with estimation of the Cohen d statistic, adjusting for the variables that may influence the results. A multilevel analysis will be performed to determine the effect of the different pilot sites or schools. The effect of the intervention could be modified by gender, cultural and socioeconomic level, body mass index (BMI), as well as by the baseline lifestyles, which will be controlled in the analysis. Separate analyses will also be performed for females, males, low and high socio-economic level to assess the effect of the intervention in these categories of interest. The level of statistical significance will be set at α=0.05 and all tests will be two-tailed. Statistical analyses will be carried out using the software packages SPSS, version 22.0 (SPSS Inc, Chicago, IL) and Stata (StataCorp. 2009. Stata Statistical Software: Release 11. College Station, TX: StataCorp LP). Conversational methods will be used to collect data in focus groups. All of them will be audio and/or videotaped and transcribed systematically, literally, and anonymously. An analysis will be made of thematic content, coding the data and grouping them into predefined categories based on topics. The analysis will be done with the support of Atlas.Ti and by triangulation of analyst.

Ethical approval has been asked to clinical research ethics committee (CEIC) of all four pilot sites: ACCORD Medical Research Ethics Committee (AMREC) in Scotland and England, IRCCS Policlinico of Milan in Lombardy and CEIC of IDIAP Jordi Gol in Catalonia. Subjects will be informed of the objectives of the project. The confidentiality of the recruited subjects and their data will be ensured in accordance with the provision of European current legislation on personal data protection: 95/46/EC EU Directive (DPD) on Data Protection and the EU 2016/679 General Data Protection Regulation.

ELIGIBILITY:
Inclusion Criteria:

The study will include:

* Female and male adolescents aged 13 to 16 years (inclusive),
* Who agree to participate and sign the informed consent along with their parents/guardian,
* Have no physical or psychological condition that would prevent understanding of and participation in the intervention,
* Are able to participate in the study for six months, and
* Have an adequate proficiency in the local language.

Exclusion Criteria:

* Those unable to use a smartphone will be excluded from the study.

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 525 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in dietary habits | Baseline and after intervention (6 months from baseline)
  Mediterranean Diet Quality Index for children and teenagers (KIDMED) questions
Change in physical activity | Baseline and after intervention (6 months from baseline)
  The Physical Activity Questionnaire for Adolescents (PAQ-A)
Change in sedentary behaviour | Baseline and after intervention (6 months from baseline)
  The Screen time-based sedentary behaviour questionnaire (SSBQ) from the HELENA study
Change in sleeping habits | Baseline and after intervention (6 months from baseline)
  Sleep Habits Survey for Adolescents (SHSA)
Change in lifestyles knowledge questionnaire | Baseline and after intervention (6 months from baseline)
  Ad hoc questionnaire on lifestyle knowledge
Change in user experience of the PEGASO system | 4 and 6 months after baseline
  Ad-hoc interviews pro-forma to assess user experience
Change in the usability of the system | 2, 4 and 6 months after baseline
  System Usability Scale (SUS questionnaire)
Change in the emotions when using the system | 4 and 6 months after baseline
  Emotional Metric Outcomes questionnaire
Change in satisfaction when using the system | 4 and 6 months after baseline
  Ad-hoc questionnaire for satisfaction
Change in dietary habits | Baseline and after intervention (6 months from baseline)
  Ad-hoc questionnaire
Change in physical activity | Baseline and after intervention (6 months from baseline)
  Ad-hoc questionnaire

SECONDARY OUTCOMES:
Self-perceived health status | Baseline and after intervention (6 months from baseline)
  One question from the SF-12
Motivation | Baseline and month 2, 4 and 6 after baseline
  Perceived Competence Scale
Habit | Continous data collection from month 1 to month 6 with data extraction at month 6 for analysis
  Self-Report Behavioural Automaticity Index (SBRAI)
Self-awareness | Continous data collection from month 1 to month 6 with data extraction at month 6 for analysis
  COM-B-Q Self-Assessment Questionnaire
Weight | Baseline and after intervention (6 months from baseline)
Height | Baseline and after intervention (6 months from baseline)
Percentage of body fat | Baseline and after intervention (6 months from baseline)
Waist circumference | Baseline and after intervention (6 months from baseline)

OTHER OUTCOMES:
Parental information (education and occupation) | Baseline
  Ad-hoc questionnaire

REFERENCES:
- [Derived] Caon M, Prinelli F, Angelini L, Carrino S, Mugellini E, Orte S, Serrano JCE, Atkinson S, Martin A, Adorni F. PEGASO e-Diary: User Engagement and Dietary Behavior Change of a Mobile Food Record for Adolescents. Front Nutr. 2022 Mar 17;9:727480. doi: 10.3389/fnut.2022.727480. eCollection 2022. PMID 35369096
- [Derived] Puigdomenech E, Martin A, Lang A, Adorni F, Gomez SF, McKinstry B, Prinelli F, Condon L, Rashid R, Caon M, Atkinson S, Lafortuna CL, Ciociola V, Hanley J, McCloughan L, Castell C, Espallargues M; PEGASO Fit For Future Consortium. Promoting healthy teenage behaviour across three European countries through the use of a novel smartphone technology platform, PEGASO fit for future: study protocol of a quasi-experimental, controlled, multi-Centre trial. BMC Med Inform Decis Mak. 2019 Dec 17;19(1):278. doi: 10.1186/s12911-019-0958-x. PMID 31847919